CLINICAL TRIAL: NCT05225454
Title: The Life Style Patterns and the Development Trend of Chronic Diseases in Healthy and Sub-healthy Groups Were Analyzed by Using Data-mining Techniques
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 110027-E
Record Dates: First submitted 2021-10-21; First posted 2022-02-04 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease Stage 1; Chronic Kidney Disease Stage 2; Chronic Kidney Disease Stage 3; Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 5; Metabolic Syndrome; Chronic Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Metabolic Syndrome; Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Used multi-year health examination member profile by multi-algorithms technology, to find comprehensive key hazard factors or important high-risk group components for metabolic syndrome and chronic kidney disease or more common chronic diseases.

DETAILED DESCRIPTION:
The proportion of the population over the age of 65 in Taiwan reached 7.10% in 1993. After Taiwan became an 「aging country」, the originally slow growth of the elderly population (9.9% in 2006) started to increase, and it reached 14.05% in 2018, which was almost 2 times that in 1993. In addition, Taiwan formally became an 「aged country」as defined globally. According to the statistical data from the Ministry of the Interior and the data from the National Development Council, it is estimated that the population over the age of 65 is rapidly growing. It is expected that 6 years later (by 2026), the elderly population in Taiwan will exceed 20%. Taiwan will formally become the「super-aged country」as defined globally, with a population structure similar to that in Japan, South Korea, Singapore, and some European countries (Department of Statistics, 2018; National Development Council, 2019). In order to effectively prevent and treat chronic diseases of sub-health populations and develop health management prediction systems that have unlimited market opportunities and potentials, the author intends to extend the achievements of individual projects sponsored by the Ministry of Science and Technology in recent years. By multi-year complete health examination member profile, this project used multiple algorithms, such as Logistic regression (LR); Classification And Regression Trees (CART); Hierarchical Linear Modeling (HLM); Random forests (RF); Support-Vector Machines (SVM); eXtreme Gradient Boosting (xGBoost); Light Gradient Boosting Machine (LightGBM) and multiple analysis tools to explore the common potential health hazard variables of the sub-health population to establish a comprehensive assessment health management system that can detect chronic diseases early, the research results will be provided for reference in related fields.

ELIGIBILITY:
Inclusion Criteria:

* Continuously health screening twice or more in MJ health reports.
* Chronic kidney disease
* Metabolic syndrome
* Or more, common chronic diseases

Exclusion Criteria:

* Participants who have received clinical treatment
* Subjects of other related research diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In 2006-2017 of the MJ Health Research Foundation's member, of the de-linked and de-identified annual health check database, about 71,108 people; 2015-2020, the Health2Sync provides [Intelligent Anti-Glucose System], the biometric and behavioral item de-linked and de-identified data, about 10,000 people.
Sampling Method: Non-Probability Sample
Enrollment: 81108 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-07-03 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with metabolic syndrome in kidney disease-related adverse events as assessed by estimated glomerular filtration rate | 2 year
  Physiological information of participants with chronic kidney disease related adverse events as assessed in metabolic syndrome, by natural longitudinal change from baseline in estimated glomerular filtration rate at 2 years recent in health screening in participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Oriental Institute of Technology / Far Eastern Memorial Hospital, New Taipei City, Pan-Chiao Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No